CLINICAL TRIAL: NCT04877301
Title: Use of Ultrasound Guidance to Facilitate Insertion of Peripheral Intravenous Catheter in Pediatric Patients
Brief Title: Use of Ultrasound Guidance to Facilitate Obtaining Peripheral Intravenous Access
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty enrolling
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIN001
Record Dates: First submitted 2012-12-11; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2013-08

CONDITIONS: Catheterization, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound guidance (Experimental): Ultrasound guidance used to facilitate insertion of PIV catheter.
  Interventions: Device: Ultrasound guidance
- Non-ultrasound guidance (Active Comparator): Ultrasound guidance will not be used for insertion of PIV catheter.
  Interventions: Procedure: Non-ultrasound guidance

INTERVENTIONS:
Device: Ultrasound guidance — Ultrasound guidance used to facilitate insertion of PIV catheter
  Arms: Ultrasound guidance
Procedure: Non-ultrasound guidance — Ultrasound guidance will not be used for insertion of PIV catheter
  Arms: Non-ultrasound guidance

SUMMARY:
The purpose of this study is to determine if the use of ultrasound guidance to insert peripheral intravenous catheters will decrease the number of punctures required to successful insertion. The hypothesis is that fewer attempts will be required with the use of ultrasound potentially leading to preservation of vessels, decreased patient pain scores and increased patient/parent satisfaction.

DETAILED DESCRIPTION:
Patients with known or current difficult venous access will be referred to the Vascular Access Team for peripheral intravenous catheter insertion. The Vascular Access Team will randomize patients to ultrasound guidance or non-ultrasound guidance for placement of the peripheral intravenous catheter.

ELIGIBILITY:
Inclusion Criteria:

* patients 0-17 years of age requiring peripheral intravenous access
* have not had PIV attempt in preceding 24 hours

Exclusion Criteria:

* patients who are medically unstable
* patients who require emergent intravenous access

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-12 (Estimated); Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Number of attempts to successful peripheral intravenous access cannulation. | 1 time - baseline visit

SECONDARY OUTCOMES:
Patient pain score rating for PIV access attempt. | 1 time - baseline visit

OTHER OUTCOMES:
Parent satisfaction with child's PIV access experience. | 1 time - baseline visit
PIV extravasations. | 1 time - baseline visit
  Cincinnati Children's Hospital has an initiative to reduce the number of PIV extravasations. The investigators will measure the number of extravasations in the study participants to determine if ultrasound guidance has an effect on this number.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon A Dwyer, ADN, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Neil Johnson, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Background] American Academy of Pediatrics Committee on Psychosocial Aspects of Child and Family Health, American Pain Society, Task Force on Pain in Infants, Children, and Adolescents (2001). The assessment and management of acute pain in infants, children, and adolescents. American Academy of Pediatrics, 108, 793-797.
- [Background] Bair AE, Rose JS, Vance CW, Andrada-Brown E, Kuppermann N. Ultrasound-assisted peripheral venous access in young children: a randomized controlled trial and pilot feasibility study. West J Emerg Med. 2008 Nov;9(4):219-24. PMID 19561750
- [Background] Clark E, Giambra BK, Hingl J, Doellman D, Tofani B, Johnson N. Reducing risk of harm from extravasation: a 3-tiered evidence-based list of pediatric peripheral intravenous infusates. J Infus Nurs. 2013 Jan-Feb;36(1):37-45. doi: 10.1097/NAN.0b013e3182798844. PMID 23271150
- [Background] Costantino TG, Parikh AK, Satz WA, Fojtik JP. Ultrasonography-guided peripheral intravenous access versus traditional approaches in patients with difficult intravenous access. Ann Emerg Med. 2005 Nov;46(5):456-61. doi: 10.1016/j.annemergmed.2004.12.026. PMID 16271677
- [Background] Doniger SJ, Ishimine P, Fox JC, Kanegaye JT. Randomized controlled trial of ultrasound-guided peripheral intravenous catheter placement versus traditional techniques in difficult-access pediatric patients. Pediatr Emerg Care. 2009 Mar;25(3):154-9. doi: 10.1097/PEC.0b013e31819a8946. PMID 19262420
- [Background] Johnstone M. The effect of lorazepam on the vasoconstriction of fear. Anaesthesia. 1976 Sep;31(7):868-72. doi: 10.1111/j.1365-2044.1976.tb11897.x. PMID 9838
- [Background] Kuensting LL, DeBoer S, Holleran R, Shultz BL, Steinmann RA, Venella J. Difficult venous access in children: taking control. J Emerg Nurs. 2009 Sep;35(5):419-24. doi: 10.1016/j.jen.2009.01.014. Epub 2009 Mar 21. No abstract available. PMID 19748021
- [Background] Sandhu NP, Sidhu DS. Mid-arm approach to basilic and cephalic vein cannulation using ultrasound guidance. Br J Anaesth. 2004 Aug;93(2):292-4. doi: 10.1093/bja/aeh179. Epub 2004 Jun 11. PMID 15194622
- [Background] Walsh, G. (2008). Difficult peripheral venous access: recognizing and managing the patient at risk. Journal of the Association for Vascular Access, 13, 198-203.
- [Background] Yen K, Riegert A, Gorelick MH. Derivation of the DIVA score: a clinical prediction rule for the identification of children with difficult intravenous access. Pediatr Emerg Care. 2008 Mar;24(3):143-7. doi: 10.1097/PEC.0b013e3181666f32. PMID 18347490